CLINICAL TRIAL: NCT01504919
Title: Reducing Cancer Disparities Among Latinos in Texas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010-0606; NCI-2012-00029 (Registry Identifier: NCI CTRP); 5U54CA153505 (NIH)
Record Dates: First submitted 2012-01-03; First posted 2012-01-06 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Psychosocial Problem
Keywords: Psychosocial; Behavioral intervention; Nicotine patch; Latinos; Mexican American; Motivation and Problem Solving; MAPS; Cancer risk reduction; Smoking cessation; Overweight/obese smokers; BMI greater than or equal to 25; Wellness program; Questionnaires; Surveys; Self-help materials; Pamphlets
MeSH Terms: conditions — Smoking Cessation; Overweight | interventions — Surveys and Questionnaires; Counseling; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Education (HE) (Experimental): HE of brief counseling and self-help materials addressing 3 risk behaviors, referrals to available resources, and a home-based exercise kit; 6-week supply of nicotine patches for smoking cessation if needed.
  Interventions: Behavioral: Health Education; Behavioral: Questionnaires; Drug: Nicotine Patches
- Motivation and Problem Solving (MAPS) (Experimental): HE counseling, self-help materials, and resource referrals, and home-based exercise kit; 6-week supply of nicotine patches for smoking cessation if needed. Plus 9 proactive, telephone counseling sessions over the 18 month period.
  Interventions: Behavioral: Health Education; Behavioral: Questionnaires; Behavioral: Telephone Counseling Sessions; Drug: Nicotine Patches

INTERVENTIONS:
Behavioral: Health Education — Brief counseling at baseline, at 6 months and again at 12 months, and self-help materials addressing smoking cessation, diet, physical activity, referrals to available resources, and a home-based exercise kit (e.g., pedometer, exercise ball, strength training cables).
Behavioral: Questionnaires — Computer-based questionnaires completed at baseline, then every 6 months taking 60-90 minutes to complete.
  Other Names: surveys
Behavioral: Telephone Counseling Sessions — 9 proactive, telephone counseling sessions over 18 months. Each of these phone calls should last about 20-30 minutes.
  Other Names: Counseling
  Arms: Motivation and Problem Solving (MAPS)
Drug: Nicotine Patches — 6-week supply of nicotine patches given to participants ready to quit smoking.

SUMMARY:
The goal of this research study is to learn if a wellness program can help improve diet and physical activity levels and encourage smoking cessation in Latino individuals who are overweight.

DETAILED DESCRIPTION:
Day 1 Study Visit:

If you are found eligible to take part in this study, the following tests and procedures will be performed on Day 1 (the same day you complete the screening tests and sign this consent form):

* You will be asked to complete some computer-based questionnaires or paper/pencil questionnaires that will include questions about your feelings, moods, and smoking status. These will take 60-90 minutes to complete.
* You will have your height, weight, and waistline measured.
* Your blood pressure will be measured by a trained research staff member
* You will complete a breath test to help researchers estimate (guess) the amount of cigarette smoke you inhale. The breath test uses a disposable cardboard tube that is attached to a machine, and you will be asked to blow a long, slow, steady breath into it.
* You will be given an accelerometer to wear for 7 days. An accelerometer is a small device that is worn on the waistline of your pants that measures your level of physical activity. After 7 days, you will be asked to "turn off" and mail back the accelerometer using a prepaid envelope provided by the study staff.
* You will give a saliva sample at this visit. To collect the saliva sample, you will place a piece of cotton in your mouth for 3 minutes. The saliva sample is used to check the amount of cotinine in the body. Cotinine is a chemical that is produced in your saliva when your body breaks down nicotine.

Study Groups and Study Procedures:

At the Day 1 study visit, you will be randomly assigned (as in the flip of a coin) into 1 of 2 study groups. There is an equal chance of being assigned to either group.

Participants in both groups will receive health education on Day 1, and again 6 and 12 months later. You can also ask to receive a 6-week supply of nicotine patches, whenever you are ready to try to quit smoking and a home-based exercise kit when you are ready to begin an exercise program.

At the Day 1 health education session, the following will take place:

* You will have a brief counseling session with a study staff member to talk about smoking, diet, and your physical activity level.
* You will be offered referrals to available resources for help with your smoking cessation, diet, and physical activity.
* You will be given a home-based exercise kit, along with self-help materials that are designed to help you learn how to quit smoking and how to improve your diet and physical activity.

At the Months 6 and 12 health education sessions, the Day 1 activities will be repeated, and the following procedures will also take place:

* You will complete a computer-based or paper/pencil questionnaire about your mood, diet, and physical activity. This will take 60-90 minutes to complete.
* Your weight and waistline will be measured.
* You will complete a breath test. The breath test uses a disposable cardboard tube that is attached to a machine, and you will be asked to blow a long, slow, steady breath into it.
* You will give a saliva sample. To collect the saliva sample, you will place a piece of cotton in your mouth for 3 minutes. The saliva sample is used to check the amount of cotinine in the body. Cotinine is a chemical that is produced in your saliva when your body breaks down nicotine.
* You will be given an accelerometer to wear for 7 days. After 7 days, you will mail back the accelerometer using a prepaid envelope provided by the study staff.

You will also have a follow-up study visit at Month 18. During this visit, the same procedures from the Month 12 visit will be performed. However, you will not have a health education session at Month 18.

Wellness Program:

In addition to the health education visits and materials, participants in Group 2 will also take part in the wellness program. For the wellness program, you will receive 18 counseling phone calls over the 18 months you are on study. Each of these phone calls should last about 20-30 minutes.

The telephone counseling sessions will be digitally recorded. Audio recordings will be erased once the data have been published. The recordings will be used to help the researchers make sure that the counselors are following the correct procedures and may be used in the future to help the researchers better understand or improve the counseling treatment. No one but the researchers and their staff will be allowed to view or listen to the recordings, and the identity of the participants will be kept strictly confidential. Your study identification number will be stated by the counselor at the beginning of the taped session. The recordings are stored digitally, encrypted, and password protected.

Questionnaire Data:

Your questionnaire data will be used for research purposes only. Your responses will not be shared with your doctor. If you feel you need a doctor's opinion about anything that is asked about in the questionnaires (such as mental or emotional difficulties or symptoms), please contact either your personal doctor or the study chair.

Length of Study:

You will remain on the study for up to 18 months. Your participation on this part of the study will be over once you complete the study visit at Month 18.

Other Important Information:

* You may be contacted by phone, mail, and/or email at any time while you are taking part in this study to be reminded about the study visits. You will be asked to give the study chair the names and contact information for family members and/or friends that the study staff can contact if they cannot reach you.
* If the accelerometer is lost or stolen, you will not be responsible for the replacement cost, but you should tell the study chair right away.

This is an investigational study. The nicotine patch is FDA approved and commercially available. Up to 500 participants overall will take part in this research study. Up to 400 participants will take part in this portion of the study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Latino adults
2. 18 years of age or older
3. Current smoker with a history of smoking an average of at least 1 cigarette per day during the last year
4. Overweight/obese (BMI greater than or equal to 25)
5. Functioning telephone number
6. Valid home address
7. Ability to engage in low to moderate physical activity as determined by the Physical Activity Readiness Questionnaire (PAR-Q)
8. Blood Pressure readings <140/90 mm Hg as defined by the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; Pressure readings >/=140/90 mm Hg will be deemed ineligible to participate and excluded from the study. They will be referred to their family physician or community services. Those ineligible based on their initial blood pressure reading are allowed to participate if they provide a letter from a physician who will continue to monitor the participant during the research study.
9. Can speak, read, and understand Spanish and/or English

Exclusion Criteria:

1. Pregnancy or lactation
2. Participants who were recruited for the pilot and focus groups are not eligible for the randomized trial.
3. Contraindication for nicotine patch use
4. Regular use of tobacco products
5. Current use of tobacco cessation medications
6. Currently enrolled in another smoking cessation study
7. Another household member enrolled in the study
8. Scores below 38 on the Short Assessment of Health Literacy for Spanish Adults (SAHLSA)
9. Active substance abuse or dependence
10. Scores below the 6th grade literacy level on the Rapid Estimate of Adult Literacy in Medicine (REALM)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Efficacy of Motivation and Problem Solving (MAPS) in Cancer Risk Reduction | 6 months
  Generalized linear mixed model regression (GLMM) used in analyzing the effects of motivation and problem solving (MAPS) on the primary outcomes across the 6, 12, and 18-month time points.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Basen-Engquist, PHD, BA, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - William Marsh Rice University, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Castro Y, Basen-Engquist K, Fernandez ME, Strong LL, Eakin EG, Resnicow K, Li Y, Wetter DW. Design of a randomized controlled trial for multiple cancer risk behaviors among Spanish-speaking Mexican-origin smokers. BMC Public Health. 2013 Mar 18;13:237. doi: 10.1186/1471-2458-13-237. PMID 23506397
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org